CLINICAL TRIAL: NCT01115556
Title: This is a Single-masked Study to Compare Intravitreally Administered 0.5 mg Ranibizumab to 2.0 mg Ranibizumab in Subjects Who Manifest Persistent or Recurrent Macular Fluid Less Than 30 Days Following Treatment With Intravitreal Anti-VEGF Therapy.
Brief Title: A Pilot Study to Evaluate the Role of High-dose Ranibizumab (2.0mg) in the Management of AMD in Patients With Persistent/Recurrent Macular Fluid Less Than 30 Days Following Treatment With Intravitreal Anti-VEGF Therapy (the LAST Study)
Acronym: LAST
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vitreous -Retina- Macula Consultants of New York (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FVF4836S
Record Dates: First submitted 2010-04-30; First posted 2010-05-04 (Estimated); Results first posted 2017-10-06 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Lucentis 2.0 mg (Experimental): Lucentis 2.0 mg
  Interventions: Drug: Ranibizumab
- LUCENTIS 0.5 mg (Active Comparator)
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — 2.0 mg
  Arms: Lucentis 2.0 mg
Drug: Ranibizumab — 0.5 mg
  Arms: LUCENTIS 0.5 mg

SUMMARY:
This is a single-masked study to compare intravitreally administered 0.5 mg ranibizumab to 2.0 mg ranibizumab in subjects who manifest persistent or recurrent macular fluid less than 30 days following treatment with intravitreal anti-VEGF therapy. Patients will be masked to their treatment assignment.

The study duration is anticipated to be 12 months and will enroll 30 subjects . Patients will be randomized 2:1 to either 2.0 mg ranibizumab or 0.5mg ranibizumab.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible if the following criteria are met:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 50 years
* Subfoveal neovascularization secondary to AMD
* Best corrected visual acuity in the study eye between 20/30 to 20/400 using an ETDRS chart
* Documentation of the presence of subretinal fluid and/or cystoid macular edema on SD-OCT less than 30 days following at least six months of anti-VEGF therapy
* Presence of fibrosis, hemorrhage, or other hypofluorescent lesions should not obscure greater than 50% of the CNV lesion

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from this study:

* Pregnancy (positive pregnancy test) or lactation
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* Participation in another simultaneous medical investigation or trial
* Prior treatment with anti-VEGF therapy in the study eye within 30 days of BSL
* Prior treatment with triamcinolone in the study eye within 6 months of BSL.
* Prior treatment with dexamethasone in the study eye within 30 days prior to BSL
* Past treatment with PDT or thermal laser in the study eye
* Intraocular surgery (including cataract surgery) in the study eye within 2 months preceding BSL
* History of vitrectomy surgery, submacular surgery, or other surgical intervention for AMD in the study eye
* Active intraocular inflammation (grade trace or above) in the study eye
* Current vitreous hemorrhage in the study eye
* History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Uncontrolled glaucoma in the study eye (defined as IOP ≥ 30 mmHg despite treatment with anti-glaucoma medication)
* History of cerebral vascular accident, myocardial infarction, transient ischemic attacks within 3 months of study enrollment.
* History of allergy to fluorescein, not amenable to treatment

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K.Bailey Freund, MD, Principal Investigator — Vitreous -Retina- Macula Consultants of New York
Locations (1):
- Vitreous Retina Macula Consultants of New York, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lucentis 2.0 mg: Lucentis (ranibizumab) 2.0 mg
- Lucentis 0.5 mg: Lucentis (ranibizumab) 0.5 mg
Period: Overall Study
Arm/Group | Lucentis 2.0 mg | Lucentis 0.5 mg
Started | 7 | 2
Completed | 7 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lucentis 2.0 mg | Lucentis 0.5 mg | Total
Number analyzed (Participants) | 7 | 2 | 9
Age, Customized [Mean (Standard Deviation); unit: years] | 80.1 (5.4) | 88.0 (0.0) | 82.0 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Visual Acuity (VA) From Baseline at Month 6
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: ETDRS Letters
Arm/Group | Lucentis 2.0 mg | Lucentis 0.5 mg
Number analyzed (Participants) | 7 | 2
ETDRS Letters | 6.1 (3.7) | 2.0 (0.0)

2. Secondary Outcome: Mean Change in Visual Acuity (VA) From Baseline at Month 12
Description: * Mean change in Visual Acuity (VA) from Baseline at Month 12
  * Mean change in central foveal thickness (RPE to ILM) as measured by SD-OCT (Spectralis HRA + OCT (Heidelberg Engineering, Heidelberg, Germany) at Months 6 and 12
  * Mean change in leakage as determined by FA at Months 6 and 12
  * Mean number of ranibizumab injections at Months 6 and 12
  * Mean time to first re-treatment following the initial 3 monthly loading doses
  * Mean duration of fluid-free interval
  * Safety and tolerability of 2.0mg using the incidence and severity of adverse events
Time Frame: one year
Measure: Mean (Standard Deviation); unit: ETDRS Letters
Arm/Group | Lucentis 2.0 mg | LUCENTIS 0.5 mg
Number analyzed (Participants) | 7 | 2
ETDRS Letters | 4.1 (4.5) | 3.0 (0.0)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Lucentis 2.0 mg | Lucentis 0.5 mg
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes